CLINICAL TRIAL: NCT02001272
Title: EWOC-1 Trial: Multicenter, Randomized Trial of Carboplatin +/- Paclitaxel in Vulnerable Elderly Patients With Stage III-IV Advanced Ovarian Cancer
Brief Title: EWOC-1 Trial: Carboplatin +/- Paclitaxel in Vulnerable Elderly Patients With Stage III-IV Advanced Ovarian Cancer
Acronym: EWOC-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-772
Record Dates: First submitted 2013-11-22; First posted 2013-12-04 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Ovarian Cancer
Keywords: Elderly; Vulnerable; Ovarian cancer; Chemotherapy
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A:Paclitaxel + Carboplatin every 3 weeks (Experimental): Patients randomized to the arm A receive 6 courses the following regimen: Paclitaxel 175 mg/m²/3 hours, I.V. and carboplatin AUC 5, I.V. every 3 weeks (1 cycle = 21 days).
  Interventions: Drug: Paclitaxel + Carboplatin every 3 weeks
- B:Carboplatin monotherapy every 3 weeks (Experimental): Patients randomized to the arm B receive 6 courses the following regimen: Carboplatin monotherapy AUC 5 or 6 every 3 weeks (1 cycle = 21 days).
  Interventions: Drug: Carboplatin monotherapy every 3 weeks
- C:Weekly Paclitaxel and Carboplatin (Experimental): Patients randomized to the arm C receive 6 courses the following regimen: weekly paclitaxel 60 mg/m²/1 hour and weekly carboplatin AUC 2 (d1, d8, d15 ; d1=d29) (1 cycle = 28 days).
  Interventions: Drug: Weekly Paclitaxel and Carboplatin

INTERVENTIONS:
Drug: Paclitaxel + Carboplatin every 3 weeks — Patients will receive a premedication of 130mg prednisolone the day before (22 pm) and the morning (7 am). A pretreatment using corticosteroids, antihistamines and H2 antagonists and setrons in accordance with local standards of care will be administered 30 minutes before Paclitaxel administration. At H0, Paclitaxel is administered at 175mg/m² in 3 hours then Carboplatin is administered at AUC 5mg/mL/min.
  Arms: A:Paclitaxel + Carboplatin every 3 weeks
Drug: Carboplatin monotherapy every 3 weeks — A pretreatment using setrons in accordance with local standards of care will be administered 30 minutes before Carboplatin at AUC 5 to 6mg/mL/min in 1 hour.
  Arms: B:Carboplatin monotherapy every 3 weeks
Drug: Weekly Paclitaxel and Carboplatin — A pretreatment using corticosteroids, antihistamines and H2 antagonists and setrons in accordance with local standards of care will be administered 30 minutes before Paclitaxel 60mg/m² in 1 hour followed by Carboplatin at AUC 2mg/mL/min in 1 hour.
  Arms: C:Weekly Paclitaxel and Carboplatin

SUMMARY:
The current standard of first-line chemotherapy in advanced ovarian cancer is the combination of carboplatin AUC 5mg/mL/min and paclitaxel 175 mg.m-². This combination is feasible in selected elderly patients such as those included in prospective trials. These trials, however, include a minority of the elderly population. In wider selection of patients >70 years old, the standard carboplatin-paclitaxel regimen has been shown to induce an excess of toxicity and premature treatment stopping. For elderly patients thought to be vulnerable and at high risk of toxicity with the standard 3-weekly carboplatin-paclitaxel regimen, other options are used in routine practice. One option is to delete paclitaxel and treat elderly patients with carboplatin as a single agent. An alternative is to use the carboplatin-paclitaxel regimen in a weekly schedule for both drugs such as reported by the MITO (Multicentre Italian Trial in Ovarian Cancer).

To date, there is no randomized trial which could give us some evidence of how to select patients who could benefit most of one or the other regimen described above. The 4th Ovarian Cancer Consensus Conference has indeed recognised the medical unmet need of adapted therapy for elderly patients with ovarian cancer and the necessity of additional research in this population.

Recently, GINECO has described a Geriatric Vulnerability Score (GVS) in a population of elderly patients with advanced ovarian cancer included in a specific multicenter phase II trial. The best proportional hazard model fitting for overall survival identified the following geriatric covariates score as being poor survival risk factors: ADL score <6, IADL score <25, HADS score >14, albuminemia <35g/L and , lymphopenia <1G/L. GVS is the sum of these risk factors for each patient. Using a cut off of 3, the GVS identified a group of patients at high risk of severe toxicity, early cessation of treatment, unplanned hospitalization and adverse outcomes.

This international multicentre randomized phase II trial will compare the success rate of delivering 6 courses of chemotherapy with evidence of efficacy and without premature termination for progression, death or unacceptable toxicity of three different chemotherapy regimens in a selected population of elderly patients with a GVS ≥ 3:

* Arm A: Paclitaxel 175mg/m²/3 hours, I.V. and carboplatin AUC 5, I.V. every 3 weeks
* Arm B: Carboplatin monotherapy AUC 5 or 6 every 3 weeks
* Arm C: Weekly paclitaxel 60 mg/m²/1 hour and weekly carboplatin AUC 2 (d1, d8, d15 every 4 weeks)

The total number of patients to be enrolled is 240, ie 22 in each arm (total = 66) at the first step, then 58 more by arm (total=174) after interim analysis.

ELIGIBILITY:
Inclusion Criteria:

* Woman >70 year old
* Histologically or cytologically proven FIGO stage III to IV epithelial ovarian cancer or peritoneal primary or fallopian tube. A cytological proof is accepted if associated with a ratio of CA125/CEA >25 and a radiological pelvic mass.
* GVS (Geriatric Vulnerability Score) >3.
* Adequate bone marrow function including the following: Neutrophils ≥ 1.5 x 109/L , platelets ≥100 x 109/L and hemoglobin ≥9 g/dL.
* Adequate glomerular filtration rate >40 ml/min (estimates based on MDRD or Chatelut formula are sufficient)
* No icterus.
* Life expectancy > 3 months.
* Written informed consent obtained.
* Covered by a Health System where applicable

Exclusion Criteria:

* Other malignancy within the last 5 years, except for adequately treated carcinoma in situ of the cervix or squamous carcinoma of the skin, or adequately controlled limited basal cell skin cancer.
* Prior history of chemotherapy.
* Prior history of radiotherapy which may affect patient tolerability to chemotherapy.
* Major perturbations of liver biology: Bilirubin > 2 fold the upper normal limit (UNL), SGOT-SGPT > 3 fold UNL.
* Patient unable to be regularly followed for any reason (geographic, familial, social, psychologic).
* Any mental or physical handicap at risk of interfering with the appropriate treatment.
* Known allergy to Cremophor ® EL -containing drugs.
* Any administrative or legal supervision where applicable

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Treatment success.Treatment success is defined as the ability to deliver 6 courses of chemotherapy without premature termination for progression, death or unacceptable toxicity | After 6 courses of chemotherapy i.e 4.5 to 6 months (depending on the arm)
  Treatment success is defined as the ability to deliver 6 courses of chemotherapy without premature termination for progression, death or unacceptable toxicity. Unacceptable toxicity is defined as a major adverse event related to chemotherapy or treatment procedure leading either to early treatment stopping, to an unplanned hospital admission or to death or to a dose delay lasting more than 14 days or more than 2 dose reductions.

SECONDARY OUTCOMES:
Therapeutical strategy | At the end of treatment (6 courses ), i.e 4.5 to 6 months (depending on the arm)
  Therapeutical strategy will be assessed by measuring the feasibility of performing an optimal surgery and feasibility of performing neoadjuvant chemotherapy and surgery and post operative chemotherapy until 6 courses in case of planned interval debulking surgery.
Overall Survival | 2.5 years
  Overall survival is defined as the time period from the date of randomization to the date of death.
Progression-free survival | 2.5 years
  Progression-free survival is defined as the time period from the date of randomization to the date of disease progression or death whichever occurs first.
Quality of Life | At the end of treatment (6 courses ), i.e 4.5 to 6 months (depending on the arm)
  Quality of life is evaluated using the FACT-O questionnaire
Safety and tolerability | At the end of treatment (6 courses ), i.e 4.5 to 6 months (depending on the arm)
  Adverse events are defined using the NCI-CTC AE scale version 4.3
Aging biomarkers | At the end of treatment (6 courses ), i.e 4.5 to 6 months (depending on the arm)
  Aging biomarkers are represented by the expression level of cathelin-related antimicrobial peptide or CRAMP, stathmin, EF-1α, and chitinase

CONTACTS AND LOCATIONS:
Overall Officials: Claire FALANDRY, MD, Principal Investigator — Service d'oncogériatrie, Centre Hospitalier Lyon Sud, Hospices Civils de Lyon
Locations (63):
- Notre-Dame Hospital of the CHUM, Montreal, Canada
- Herlev Hospital, Herlev, Denmark
- Kuopio University Hospital, Kuopio, Finland
- France (53):
  - Service d'Oncologie Médicale - Centre Hospitalier d'Alès, Alès
  - Service d'Oncologie Médicale - ICO Paul Papin, Angers
  - Service de cancérologie clinique - Institut Sainte-Catherine, Avignon
  - Servide d'Oncologie Médicale - Hôpital Jean Minjoz, Besançon
  - Service d'Oncologie Médicale - Institut Bergonié, Bordeaux
  - Service d'Onco-Hématologie - Hôpital Fleyriat, Bourg-en-Bresse
  - Service de Radiothérapie et Oncologie Médicale - Hôpital Morvan, Brest
  - Service d'Uro-Gynécologie - Centre François Baclesse, Caen
  - Service d'Oncologie - Centre Hospitalier de Chambéry, Chambéry
  - Service d'Oncologie Médicale - Centre Hospitalier de Cholet, Cholet
  - Servide d'Oncologie Médicale - Centre Jean Perrin, Clermont-Ferrand
  - Service d'Oncologie - Centre Hospitalier Alpes Leman, Contamines Sur Arve
  - Service d'Oncologie Radiothérapie - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Service d'Oncologie Médicale - Centre d'Oncologie et de Radiothérapie du Parc, Dijon
  - Service d'Oncologie Médicale - Centre Georges François Leclerc, Dijon
  - Service de Médecine Gériatrique - Centre Hospitalier Intercommunal des Alpes du Sud -Site de Gap, Gap
  - Service d'Oncologie Médicale - Hôpital Michallon - CHU Grenoble, Grenoble
  - Service d''Hématologie Oncologie - Hôpital André Mignot, Le Chesnay
  - Service d'Oncologie Médicale - Centre Jean Bernard - Clinique Victor Hugo, Le Mans
  - Service de Médecine Interne et Oncologie Médicale - CH du Mans, Le Mans
  - Service d'Oncologie - Hôpital Dupuytren, Limoges
  - Service d'Oncologie Service 2 B Nord - Centre Léon Bérard, Lyon
  - Service d'Oncologie Médicale - Institut Paoli Calmettes, Marseille
  - Service d'Oncologie multidisciplinaire - Hôpital Nord, Marseille
  - Service d'Oncologie Médicale - Institut Régional du Cancer Montpellier, Val d'Aurelle, Montpellier
  - Service d'Oncologie Médicale - Centre Azuréen de Cancérologie, Mougins
  - Service de Chimiothérapie - Centre Catherine de Sienne, Nantes
  - Service d'Onco-Hématologie - Centre Antoine Lacassagne, Nice
  - Service d'Oncologie Radiothérapie - Clinique de Valdegour, Nîmes
  - Servicde d'Oncologie Médicale - Centre Hospitalier Régional d'Orléans, Orléans
  - Service d'Oncologie Médicale - Hôpital des Diaconesses, Paris
  - Service d'Oncologie - Hôpital Cochin, Paris
  - Service d'Oncologie - Groupe Hospitalier Saint-Joseph, Paris
  - Service d'Oncologie Médicale - Hôpital Européen Georges Pompidou, Paris
  - Service d'Oncologie Médicale - Centre Hospitalier de Perpignan, Perpignan
  - Service oncogériatrie, Centre Hospitalier Lyon Sud, Hospices Civils de Lyon, Pierre-Bénite
  - Centre CARIO - Hôpital Privé des Côtes d'Armor, Plerin Sur Mer
  - Servide d'Oncologie Médicale - Centre Hospitalier de la Région d'Annecy, Pringy
  - Servide de Radiothérapie et Oncologie Médicale - Centre Hospitalier Intercommunal de Cornouaille, Quimper
  - Servide d'Oncologie Médicale - Institut Jean Godinot, Reims
  - Service d'Oncologie Médicale - Centre Hospitalier Yves le Foll, Saint-Brieuc
  - Service d'Oncologie Radiothérapie - Centre Hospitalier Privé de Saint-Grégoire, Saint-Grégoire
  - Service d'Oncologie Médicale - ICO Centre René Gauducheau, Saint-Herblain
  - Service de Médecine interne et oncologie - Hôpital Inter Armées de Begin, Saint-Mandé
  - Service d'Oncologie Médicale - Clinique Mutualiste de l'Estuaire, Cité Sanitaire, Saint-Nazaire
  - Service d'Oncologie Médicale - Groupe Hospitalier Public du Sud de l'Oise - Site de Senlis, Senlis
  - Service d'Oncologie Médicale - Centre Hospitalier de Sens, Sens
  - service d'Oncologie Médicale - Centre Hospitalier Broussais, St-Malo
  - Service d'Oncologie Médicale - Centre Paul Strauss, Strasbourg
  - Service de Chirurgie et Oncologie Gynécologique et Mammaire - Hôpitaux du Léman, Thonon-les-Bains
  - Service d'Oncologie Médicale - Institut Claudius Regaud, Toulouse
  - Service d'Oncologie Médicale - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Service de Médecine Oncologique - Institut de Cancérologie Gustave Roussy, Villejuif
- Italy (6):
  - Centro di Riferimento Oncologico - CRO,IRCCS, Aviano
  - Azienda Ulss 21 Legnago, Legnago
  - Fondazione IRCCS Istituto Nazionale Tumori, Milan
  - Ulls13 - Mirano, Mirano
  - Ospedale Nuovo di Sassuolo, Sassuolo
  - Fondazione del Piemonte per l'Oncologia - Istituto di Candiolo, Torino
- Linköping University Hospital, Linköping, Sweden

REFERENCES:
- [Result] Falandry C, Rousseau F, Mouret-Reynier MA, Tinquaut F, Lorusso D, Herrstedt J, Savoye AM, Stefani L, Bourbouloux E, Sverdlin R, D'Hondt V, Lortholary A, Brachet PE, Zannetti A, Malaurie E, Venat-Bouvet L, Tredan O, Mourey L, Pujade-Lauraine E, Freyer G; Groupe d'Investigateurs Nationaux pour l'Etude des Cancers de l'Ovaire et du sein (GINECO). Efficacy and Safety of First-line Single-Agent Carboplatin vs Carboplatin Plus Paclitaxel for Vulnerable Older Adult Women With Ovarian Cancer: A GINECO/GCIG Randomized Clinical Trial. JAMA Oncol. 2021 Jun 1;7(6):853-861. doi: 10.1001/jamaoncol.2021.0696. PMID 33885718
- [Result] Falandry C, Pommeret F, Gladieff L, Tinquaut F, Lorusso D, Mouret-Reynier MA, D'Hondt V, Mollon-Grange D, Floquet A, Abadie-Lacourtoisie S, Brachet PE, Stefani L, Rousseau F, Frenel JS, Del Piano F, Komulainen M, Warkus T, Tredan O, Pujade-Lauraine E, Freyer G. Validation of the geriatric vulnerability score in older patients with ovarian cancer: an analysis from the GCIG-ENGOT-GINECO EWOC-1 study. Lancet Healthy Longev. 2022 Mar;3(3):e176-e185. doi: 10.1016/S2666-7568(22)00002-2. Epub 2022 Feb 4. PMID 36098291
- See also: Related Info — http://www.arcagy.org
- See also: Related Info — http://www.esgo.org/engot/Pages/AboutENGOT.aspx